CLINICAL TRIAL: NCT05807308
Title: Technology-Based Cognitive and Artistic Therapeutic Activities
Brief Title: The Effect of Technology-Based Cognitive and Artistic Therapeutic Activities on the Mental Status of Children With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Çiğdem Sarı Öztürk, Gazi University, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CSOZTURK-15/03
Record Dates: First submitted 2023-03-15; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Children Followed up With Cancer Diagnosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- technology-based cognitive and artistic therapeutic activities (Experimental): The group receiving technology-based cognitive and artistic therapeutic activities
  Interventions: Behavioral: Technology-based cognitive and artistic therapeutic activities
- Control group (No Intervention): the group that did not receive any training

INTERVENTIONS:
Behavioral: Technology-based cognitive and artistic therapeutic activities — Therapeutic and artistic activities within the program (drawing, mandala, etc.). The program will be implemented in 6 sessions in two weeks. At the beginning and end of the program, children's anxiety and spiritual well-being levels will be evaluated.
  Arms: technology-based cognitive and artistic therapeutic activities

SUMMARY:
This research will be carried out to determine the effects of technology-based cognitive and artistic therapeutic activities on the mental state of children receiving cancer treatment. The research will be conducted in a single-blind parallel group randomized controlled trial design. A program consisting of six two-week sessions will be implemented. The program will include many artistic activities such as therapeutic and drawing.

DETAILED DESCRIPTION:
In the study, a program consisting of technology-based cognitive and artistic activities will be applied to children followed up with cancer diagnosis. Therapeutic and artistic activities within the program (drawing, mandala, etc.). The program will be implemented in 6 sessions in two weeks. At the beginning and end of the program, children's anxiety and spiritual well-being levels will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 9-18,
* Those receiving cancer treatment,
* At least two months have passed since the start of treatment,
* Those who have internet access on their smartphone or computer

Exclusion Criteria:

* Those who have experienced an important life event other than illness (parents' divorce, death, moving, etc.) in the last six months,
* Those who have not received chemotherapy treatment,
* In the terminal period,
* Children with a severe psychological diagnosis

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Spielberger State-Trait Anxiety Inventory for children | Change from Baseline level of Spielberger State-Trait Anxiety to 2 weeks (change is being assessed)
  The scale is a 20-item self-report measure of anxiety using a 4-point Likert-type scale (from 0 to 3 points) for each item. The total score obtained from the scale varies between 20 and 60. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Adolescent Spiritual Well-Being Scale | Change from Baseline level of Adolescent Spiritual Well-Being Scale to 2 weeks (change is being assessed)
  The scale is a 34-item self-report measure of anxiety using a 5-point Likert-type scale (from 0 to 3 points). The total score obtained from the scale varies between 0 and 100. The higher the score obtained from the scale, the better the spiritual well-being is determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided